CLINICAL TRIAL: NCT01760434
Title: Prospective Study: Long-Term Pulmonary Function, Health-Related Quality of Life, and Sagittal Plane Alignment Following the Treatment of Pediatric Scoliosis
Brief Title: Long-Term Outcome Following the Treatment of Pediatric Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Scoliosis Research Society (Other)
Responsible Party: Principal Investigator, A. Noelle Larson, Co-Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-008308
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: scoliosis; long-term outcomes; sagittal plane; quality of life; curve progression; pulmonary function
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Long-Term Outcomes (Other): Patients will be recruited who were diagnosed with adolescent idiopathic scoliosis prior to age 18 and before 1994 (minimum 20 year outcomes) with available xrays. Patients will be included who were treated with surgery, observation, or bracing. Patients will return for a one-time visit for new xrays, physical exam, health-related quality of life surveys, and pulmonary function testing.
  Interventions: Other: Long-term outcomes

INTERVENTIONS:
Other: Long-term outcomes — Patients with a history of adolescent idiopathic scoliosis will return at a minimum of 20 year follow-up for new spine xrays, clinical exam, pulmonary function testing, and assessment of health related quality of life based on survey responses.

SUMMARY:
Evaluate the long-term outcomes following operative and nonoperative treatment of childhood scoliosis.

DETAILED DESCRIPTION:
The investigators hypothesize that sagittal alignment and thoracic volumes will predict successful treatment outcomes as measured by improved pulmonary function and health-related quality of life in adolescent idiopathic scoliosis patients at a minimum 20-year follow-up. Significant focus has been placed on the coronal plane in order to determine treatment indications for scoliosis, but with new understanding about the important of sagittal balance and pulmonary function, the treatment indications should be broadened. Thus, the investigators propose the following study to explore parameters associated with a durable and acceptable outcome following scoliosis treatment, minimizing the need for further surgery and to optimizing quality of life and pulmonary health. Beyond the standard radiographs and Scoliosis Research Society (SRS) scores, this study undertakes a comprehensive assessment of health-related quality of life, chest asymmetry and body satisfaction scoring, sagittal plane parameters, and 3D modeling of the childhood and current spinothoracic deformity. Thus, the investigators research team is uniquely poised to determine broader treatment indications for scoliosis. The overarching goal of this research effort is to determine new parameters based on thoracic volume and sagittal plane alignment in addition to coronal deformity in order to determine the appropriate treatment threshold for surgical intervention in children with adolescent idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adolescent idiopathic scoliosis made before age 18
* Diagnosis of adolescent idiopathic scoliosis prior to 1994
* Treatment with bracing, observation, or surgery prior to age 18 and 1994
* Adequate radiographs/medical records available from time of diagnosis

Exclusion Criteria:

* Neuromuscular scoliosis
* Syrinx
* Inadequate radiographs/medical records available from time of diagnosis

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cobb angle and sagittal plane alignment | 20 years
  Cobb angle and sagittal plane alignment at minimum 20 year follow-up after bracing, surgery or observation for adolescent idiopathic scoliosis
Scoliosis curve magnitude | Nov. 2014

SECONDARY OUTCOMES:
Pulmonary function testing | 20 years
  Pulmonary function testing will be performed at 20 years following bracing, observation or surgery for scoliosis to assess association between coronal and sagittal plane alignment and pulmonary function.
Health-related quality of life | Nov. 2014

CONTACTS AND LOCATIONS:
Overall Officials: Annalise Noelle Larson, MD, Principal Investigator — Mayo Clinic; Michael J. Yaszemski, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials